CLINICAL TRIAL: NCT04317339
Title: A Randomized，Double-blinded, Placebo-controlled Trial Evaluating the Efficacy and Safety of Zhigancao Tang Granule for HFpEF of Qi-Yin Dificiency
Brief Title: The Efficacy and Safety of Zhigancao Tang Granule for HFpEF of Qi-Yin Dificiency
Acronym: HFpEF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZGCT
Record Dates: First submitted 2020-03-04; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: heart failure with preserved ejection fraction; Qi-Yin deficiency syndrome; randomized, double blinded and controlled trial; Zhigancao Tang granule

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zhigancao Tang granule group (Experimental): Participants in experimental group will receive Zhigancao Tang granule therapy for 12 weeks. In addition, participants will receive standard heart failure treatment，including ACEI/ARB/ARNI, aldosterone antagonists, beta blockers, nitrate esters, diuretics as needed.
  Interventions: Drug: Zhigancao Tang granule
- Zhigancao Tang placebo group (Placebo Comparator): Participants in experimental group will receive Zhigancao Tang placebo granule therapy for 12 weeks. In addition, participants will receive standard heart failure treatment，including ACEI/ARB/ARNI, aldosterone antagonists, beta blockers, nitrate esters and diuretics as needed.
  Interventions: Drug: Zhigancao Tang placebo granule

INTERVENTIONS:
Drug: Zhigancao Tang granule — Zhigancao Tang: Dissolve Zhigancao Tang granule in 200ml hot water, twice a day,12 weeks, oral.
  Standard heart failure treatment，including ACEI/ARB/ARNI, aldosterone antagonists, beta blockers, nitrate esters and diuretics as needed.
  Other Names: Zhigancao Tang group; Zhigancao Tang granule group
  Arms: Zhigancao Tang granule group
Drug: Zhigancao Tang placebo granule — Zhigancao Tang placebo: Dissolve Zhigancao Tang placebo granule in 200ml hot water, twice a day,12 weeks, oral.
  Standard heart failure treatment，including ACEI/ARB/ARNI, aldosterone antagonists, beta blockers, nitrate esters and diuretics as needed.
  Other Names: Zhigancao Tang placebo group; Zhigancao Tang placebo granule group
  Arms: Zhigancao Tang placebo group

SUMMARY:
This study was designed as a randomized, double blinded and placebo-controlled clinical trial. The aim of the study is to evaluate the efficacy and safety of Zhigancao Tang granule in patients with HFpEF of Qi-Yin dificiency.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFPEF) is a clinical syndrome characterized by diastolic dysfunction.The incidence of HFpEF is increasing in recent years. Standard treatment of heart failure does not improve the prognosis of HFPEF patients. Zhigancao Tang was used to improve the symptoms of chronic heart failure in China.This randomized,double-blinded and placebo-controlled trial will objectively and standardly evaluate the effectiveness and safety of Zhigancao Tang granule.After 12 weeks of treatment, 122 HFpEF patients with deficiency of Qi and Yin were observed and evaluated in terms of heart function, clinical symptoms,exercise tolerance and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Comply with the diagnostic criteria of Western medicine for HFpEF and the diagnostic criteria for TCM syndromes of Qi-Yin deficiency;
2. Cardiac function classification by NYHA: grade I to III;
3. Age between 30 and 80 years old;
4. Those who volunteer to participate in clinical trial observation, sign informed consent and indicate date;
5. During the observation period, those who do not take other drugs other than those specified and can insist on completing the treatment and observation.

Exclusion Criteria:

1. Valvular heart disease, restrictive cardiomyopathy, pericardial disease;
2. Decompensated heart failure is unstable after treatment;
3. Combined with atrial fibrillation;
4. Patients with severe lung, liver, endocrine system and kidney dysfunction;
5. Patients with cancer and other common malignant diseases reducing life expectancy;
6. Pregnant or lactating women;
7. Allergic constitution or allergic history to common drugs;
8. Patients with mental illness or poor compliance of traditional Chinese medicine treatment.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2020-03-20 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac Functional Grading | 12 weeks
  Significant effect: cardiac function recovered to level 1 or increased by level 2; Effective: cardiac function increased by level 1 but failed to reach level 2; Ineffective: cardiac function did not change; Worsening: cardiac function decreased by level 1 or above.

SECONDARY OUTCOMES:
Ultrasonic cardiogram | 12 weeks
  Echocardiographic measurement of Left ventricular ejection fraction (LVEF), left ventricular end diastolic diameter (LVEDd), left ventricular end systolic diameter (LVESD), ratio of left ventricular early diastolic fast filling peak to late diastolic filling peak (E / a), ratio of early diastolic velocity of mitral valve to early diastolic annular velocity (E / E ').
6-min walking test (6mwt) | 12 weeks
  6 minute walking test (6mwt) is a measure of the distance the patient can reach as far as possible by walking on a hard ground without obstacles within six minutes at the fastest possible speed. It provides a comprehensive assessment of exercise capacity.
Minnesota Heart Failure Quality of Life Scale | 12 weeks
  Minnesota Heart Failure Quality of Life Scale was used to assess the impact of heart failure on life in the last four weeks. A total of 21 questions related to physical and emotional change. Higher scores mean a worse outcome.
N-terminal pro-B-type natriuretic peptide（NT-proBNP） | 12 weeks
  NT-proBNP is a reliable and sensitive indicator of heart failure. Its elevation is positively correlated with severity of heart failure.
TCM syndrome score | 12 weeks
  TCM syndrome score is used to assess changes in Qi-Yin Dificiency related symptoms during treatment. The higher the scores, the more heart failure symptoms. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Deng, M.D, Study Director — Shanghai Longhua Hospital
Locations (1):
- Longhua Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang N, Zhao Y, Liu Y, Tang N, Zheng W, Mao M, Liu Q, Shen L, Deng B. A double-blinded, placebo-controlled randomized trial evaluating the efficacy and safety of Zhigancao Tang granules for treating HFpEF: study protocol for a randomized controlled trial. Trials. 2021 Apr 20;22(1):293. doi: 10.1186/s13063-021-05232-6. PMID 33879223